CLINICAL TRIAL: NCT06939010
Title: 3D Interlocking Miniplates Versus Conventional Miniplates in Fixation of Mandibular Fractures in the Mental Foramen Region: A Split-mouth Study
Brief Title: 3D Interlocking Miniplates in Fixation of Mandibular Fractures in the Mental Foramen Region: A Split-mouth Study
Acronym: Interlocking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D-Interlocking
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Mandibular Fractures; Miniplate
Keywords: Mental nerve; conventional miniplates; 3D Interlocking; mandibular parasymphyseal fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Investigator
Masking Description: Fracture sides were allocated in a 1:1 ratio using an on-site computer software system with concealed allocation through sequentially numbered, opaque, sealed envelopes (SNOSE). Group A was treated with 3D-interlocking miniplate in one side, and Group B with conventional double miniplates configration in the other side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with bilateral fracture in the mental nerve region managed with 3D-interlocking miniplate (Experimental): patient with bilateral fracture in the mental nerve region. one side will be randomly allocated to be managed with 3D-interlocking miniplate
  Interventions: Device: 3d-interlocking miniplate
- patient with bilateral fracture in the mental nerve region managed with conventional miniplates (Experimental): patient with bilateral fracture in the mental nerve region. one side will be randomly allocated to be managed with conventional miniplates
  Interventions: Device: Conventional miniplates

INTERVENTIONS:
Device: 3d-interlocking miniplate — 3d-interlocking miniplate
  Arms: patient with bilateral fracture in the mental nerve region managed with 3D-interlocking miniplate
Device: Conventional miniplates — double miniplates in the conventional configuration
  Arms: patient with bilateral fracture in the mental nerve region managed with conventional miniplates

SUMMARY:
the study aims to compare 3D Interlocking miniplates with conventional miniplates in management of mandibular parasymphyseal fractures both clinically and radiographically.

DETAILED DESCRIPTION:
A total of 12 patients with recent bilateral parasymphyseal mandibular fractures were treated with 3D Interlocking miniplates on one side and with conventional two miniplates in the other side. Clinical evaluations were carried at multiple intervals up to 6 weeks postoperatively, with radiographic assessments performed immediately after surgery and at 12 weeks to measure mean bone density at the fracture line

ELIGIBILITY:
Inclusion Criteria:

* patients with recent bilateral mandibular fracture located in the mental foramina region.
* adults without gender predilection who agreed to follow-up,
* fractures requiring open reduction and internal fixation, and
* those medically fit for general anesthesia were included

Exclusion Criteria:

* medically compromised patients,
* fractures with infection,
* pathological or old fractures,
* completely edentulous patients,
* comminuted fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation for the assessment of mean bone density at the fracture line | 12 weeks
  Mean bone density at the fracture line was assessed using Cone-Beam Computed Tomography (CBCT) scan in Hounsfield Units (HU)

SECONDARY OUTCOMES:
Clinical evaluation for Intra-fragmentary mobility | 6 weeks
  Intra-fragmentary mobility was evaluated by bimanual palpation at the fracture site

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP